CLINICAL TRIAL: NCT01399996
Title: Influence of a Delivery System on the Efficacy of a Probiotic Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PKE PROBIOTIC
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Delayed Transit Time; Irregular Bowel Function
Keywords: probiotic; microbiota; transit time; immunity; immune function; constipation; bowel function
MeSH Terms: conditions — Constipation | interventions — Probiotics; Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Yogurt smoothie without probiotic. (Placebo Comparator)
  Interventions: Dietary Supplement: Yogurt smoothie without probiotic
- Probiotic added post fermentation. (Experimental)
  Interventions: Dietary Supplement: Yogurt smoothie with probiotic added post fermentation
- Probiotic added pre-fermentation. (Experimental)
  Interventions: Dietary Supplement: Yogurt smoothie with probiotic added pre-fermentation
- A capsule containing the probiotic. (Experimental)
  Interventions: Dietary Supplement: A capsule containing the probiotic

INTERVENTIONS:
Dietary Supplement: Yogurt smoothie without probiotic — A daily 8 oz (240 mg) serving will provide 10x^y5 cfu/ml of the probiotic (Bifidobacterium animalis subsp. lactis BB12).
  Other Names: Yogurt
  Arms: Yogurt smoothie without probiotic.
Dietary Supplement: Yogurt smoothie with probiotic added post fermentation — A daily 8 oz (240 mg) serving will provide 10x^y5 cfu/ml of the probiotic (Bifidobacterium animalis subsp. lactis BB12).
  Other Names: Yogurt with probiotic
  Arms: Probiotic added post fermentation.
Dietary Supplement: Yogurt smoothie with probiotic added pre-fermentation — A daily 8 oz (240 mg) serving will provide 10x^y5 cfu/ml of the probiotic (Bifidobacterium animalis subsp. lactis BB12).
  Other Names: Yogurt with probiotic
  Arms: Probiotic added pre-fermentation.
Dietary Supplement: A capsule containing the probiotic — A capsule taken daily will provide between 10x^y9 and 10x^y10 cfu/ml of the probiotic (Bifidobacterium animalis subsp. lactis BB12).
  Other Names: Probiotic capsule
  Arms: A capsule containing the probiotic.

SUMMARY:
In the proposed work we will evaluate the efficacy of a probiotic bacterium (Bifidobacterium animalis subsp. lactis BB12) delivered in a yogurt smoothie (organism to be added before or after fermentation) or as a supplement (tablet) by assessing 1) bowel habits (transit time); 2) the ecology of the bacterial community in the GIT; and 3) immune status of healthy human volunteers. In addition to providing information about the relative efficacy of the delivery vehicles on probiotic function it will provide novel information about the influence of the yogurt smoothie alone (control) on all the parameters measured.

DETAILED DESCRIPTION:
Probiotics (health-promoting bacteria) are often considered "functional ingredients" that act independently of the matrix used to deliver them to the human host. This thinking ignores the impact the delivery matrix (food or dietary supplement) may have on both the physiology of the probiotic organism and on the human host and is likely not true.

Historically the most common "probiotic foods" have been fermented dairy products, particularly yogurts. Since yogurts are commonly understood to contain live "good" bacteria they are well accepted by consumers. However, increasingly over the last decade, probiotics are being added to non-dairy-based foods (juice, chocolate, cookies, etc) or consumed as supplements (tablets/capsules). While this expands the options for people to obtain probiotic organism, it is not clear whether probiotics delivered in these products are as efficacious as when delivered in a dairy food. In fact, the buffering capacity and nutrient composition of milk products may directly influence efficacy of the probiotic by increasing survival during passage through the gastrointestinal tract (GIT) and by modifying the physiology of the probiotic organism. In addition, fermentation products produced by the probiotic during manufacture of yogurt may also have an influence on the efficacy of probiotic bacteria.

Our hypotheses are:

1. The vehicle used to deliver probiotic bacteria into the body influences the performance of the probiotic in vivo. Specifically, consumption of yogurt-based smoothie containing probiotic bacteria will result in greater decrease in fecal transit time, and have a greater effect on the composition of the fecal microbiota and on markers of immune status than the same probiotic bacteria delivered at the same level in the form of a dietary supplement (tablet).
2. Timing of the addition of probiotic organism to the yogurt smoothie (pre or post fermentation) will not change the efficacy of the probiotic with respect to the outcomes being assessed.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Men and women
* 18-40 years of age
* Body mass index between 20 and 35 kg/m^2
* Persons with irregular bowel function as determined using the Rome III criteria (1) which is used to classify functional gastrointestinal disorders.
* Increased gastrointestinal transit time > 60 hours.

Exclusion Criteria:

* Smoking and/or use of other tobacco products
* Blood pressure greater than 140/90 mm Hg
* A history of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease and thyroid disease (unless controlled by medication and blood results within the previous 6 months are provided).
* Lactation, pregnancy or desire to become pregnant during the study
* Use of cholesterol-lowering medication
* Refusal to discontinue intake of putative cholesterol-lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, phytoestrogens, stanol/sterol supplemented foods
* Refusal to discontinue probiotics,nutritional supplements, herbs or vitamins
* Vegetarianism/Veganism
* Lactose intolerance
* Clinical diagnosis of Inflammatory Bowel Disease (IBD), e.g. Crohn's Disease or ulcerative colitis
* Excessive alcohol consumption (> 14 standard drinks per week)
* Chronic use of anti-inflammatory medications (unless able to discontinue)
* Individuals taking stool softeners or enemas on a regular basis.
* Allergy to polyvinyl chloride (PVC) or any other type of plastic
* Individuals with a bowel transit time of < 60 hours at time of screening
* Individuals with swallowing disorders or dysphagia to food or pills
* Suspected strictures, fistulas, or physiological GI Obstruction
* GI surgery within the past three months
* Refusal to agree to give blood or plasma for the length of the study.

Note: If a participant experiences a delay in passing the capsule (beyond five days) they will be treated accordingly and excluded from future participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal transit time | Weeks 4, 10, 16, 22
  Gastrointestinal transit time is the amount of time it takes for food to travel through the digestive tract to be excreted. It will be measured using the SmartPill wireless motility capsule.

SECONDARY OUTCOMES:
Change from baseline in the fecal microbiota profile at 4 weeks following each of the 4 interventions and 1 free living period | Weeks 4, 10, 16, 22 and 28
Change from baseline in immune status at 4 weeks following each of the 4 interventions and 1 free living period | Weeks 4, 10, 16, 22, 28

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Drossman DA, Dumitrascu DL. Rome III: New standard for functional gastrointestinal disorders. J Gastrointestin Liver Dis. 2006 Sep;15(3):237-41. PMID 17013448
- [Derived] Ba Z, Lee Y, Meng H, Kris-Etherton PM, Rogers CJ, Lewis ZT, Mills DA, Furumoto EJ, Rolon ML, Fleming JA, Roberts RF. Matrix Effects on the Delivery Efficacy of Bifidobacterium animalis subsp. lactis BB-12 on Fecal Microbiota, Gut Transit Time, and Short-Chain Fatty Acids in Healthy Young Adults. mSphere. 2021 Aug 25;6(4):e0008421. doi: 10.1128/mSphere.00084-21. Epub 2021 Jul 7. PMID 34232082
- [Derived] Lee Y, Ba Z, Roberts RF, Rogers CJ, Fleming JA, Meng H, Furumoto EJ, Kris-Etherton PM. Effects of Bifidobacterium animalis subsp. lactis BB-12(R) on the lipid/lipoprotein profile and short chain fatty acids in healthy young adults: a randomized controlled trial. Nutr J. 2017 Jun 29;16(1):39. doi: 10.1186/s12937-017-0261-6. PMID 28662676
- [Derived] Meng H, Lee Y, Ba Z, Peng J, Lin J, Boyer AS, Fleming JA, Furumoto EJ, Roberts RF, Kris-Etherton PM, Rogers CJ. Consumption of Bifidobacterium animalis subsp. lactis BB-12 impacts upper respiratory tract infection and the function of NK and T cells in healthy adults. Mol Nutr Food Res. 2016 May;60(5):1161-71. doi: 10.1002/mnfr.201500665. Epub 2016 Mar 1. PMID 26821116